CLINICAL TRIAL: NCT04924257
Title: Electroconvulsive Therapy vs. Esketamine Nasal Spray in Treatment-resistant Depression: a Longitudinal, Randomized Efficacy Comparison Pilot Study
Brief Title: ECT vs. Esketamine
Acronym: ETES
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: No eligible participants
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1417/2020
Record Dates: First submitted 2021-06-07; First posted 2021-06-11 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2021-06

CONDITIONS: Treatment Resistant Depression; Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depressive Disorder, Major | interventions — Electroconvulsive Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intranasal Esketamine (Experimental)
  Interventions: Drug: Esketamine nasal spray
- ECT (Active Comparator)
  Interventions: Procedure: Electroconvulsive therapy

INTERVENTIONS:
Drug: Esketamine nasal spray — Patients will receive two treatments per week for four weeks (maximum of eight treatment sessions) or until clinical remission (MADRS <10).
  Arms: Intranasal Esketamine
Procedure: Electroconvulsive therapy — Patients will receive three treatments per week for four weeks (maximum of 12 ECT treatments) or until clinical remission (MADRS <10).
  Other Names: ECT
  Arms: ECT

SUMMARY:
Treatment-resistant depression (TRD) is a common cause of disability and one of the most common psychiatric disorders worldwide.

Electroconvulsive therapy (ECT) is currently the most effective treatment for TRD. Recent developments showed esketamine to be a rapid-acting and effective antidepressant drug and it has been hailed as a breakthrough in treating TRD. Common treatment algorithms for TRD list ECT as a treatment option, but esketamine has not yet found its exact position in those algorithms.

To the investigators' knowledge, a longitudinal, randomized controlled trial comparing the efficacy of ECT and intranasal esketamine in TRD patients has not been conducted. Furthermore, the investigators intend to measure effects of ECT and intranasal esketamine on brain connectivity and structure, using functional magnetic resonance imaging (fMRI).

In this study, inpatients with TRD at the University Hospital for Psychiatry I, Medical University Innsbruck, will be randomized to ECT or intranasal esketamine. Short- and medium-term treatment effects on functional and structural connectivity in the brain will be determined using fMRI.

ELIGIBILITY:
Inclusion Criteria:

1. DSM-5 diagnosis of Major Depressive Disorder (MDD) without psychotic features (296.22, 296.23, 296.32, 296.33) made through the Structured Clinical Interview for the DSM-V (SCID-V).
2. MADRS score ≥ 25
3. Pharmacologically treatment-resistant depressive episode [Stage ≥ II, defined by Thase & Rush (1997): failure of at least 2 adequate trials of at least 2 distinctly different classes of antidepressants (≥ 4 weeks each)] (88).
4. Age: 18 - 50 years
5. Written informed consent

Exclusion Criteria:

1. Participation in another interventional clinical trial
2. Relative contraindications to ECT treatment in accordance with the consensus paper of the Austrian Society of Psychiatry and Psychotherapy:
3. Patients who meet any exclusion criteria for nasal esketamine treatment as described in the clinical guidelines
4. Contraindications to the conduction of MRI
5. History of one or more of the following diagnoses (DSM-5):

   * MDD, single or recurrent episode with psychotic features (296.24; 296.34)
   * past or current substance dependence (except caffeine, nicotine) (303.x, 304.x, 305.x)
   * neurodevelopmental disorders (299.x, 307.x, 314.x, 315.x, 319.x)
   * schizophrenia spectrum and other psychotic disorders (293.x, 295.x, 297.x, 298.x)
   * neurocognitive disorders (290.x, 292.x, 294.x, 331.x).
6. history of ECT (unsuccessful or successful)
7. suicidal tendency requiring admission in a locked ward
8. pregnancy or lactation period
9. lack of anesthetic clearance for any other reason
10. insufficient command of German language.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
MADRS score | 4 weeks
  Reduction of Montgomery-Asberg Depression Rating Scale (MADRS, 0-60 pts.); higher score indicates more depressive symptoms; response to treatment is defined as >50% reduction in score

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Innsbruck, Innsbruck, Tyrol, Austria